CLINICAL TRIAL: NCT00135304
Title: ACHIEVE: Optimizing the Treatment of Secondary Hyperparathyroidism: A Comparison of Sensipar® and Low Dose Vitamin D vs. Escalating Doses of Vitamin D Alone
Brief Title: ACHIEVE: Optimizing the Treatment of Secondary Hyperparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050102
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Vitamin D; Sensipar®; Cinacalcet HCl; Chronic Kidney Disease
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic | interventions — Cinacalcet; Vitamin D; paricalcitol; 1 alpha-hydroxyergocalciferol

ARMS (2):
- Cinacalcet and low-dose Vitamin D (Experimental): Cinacalcet and low-dose IV Vitamin D
  Interventions: Drug: Sensipar®; Drug: Vitamin D
- Vitamin D alone (Active Comparator): Escalating doses of IV Vitamin D alone
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Sensipar® — Cinacalcet hydrochloride
  Other Names: Cinacalcet hydrochloride, Cinacalcet HCL, Cinacalcet
  Arms: Cinacalcet and low-dose Vitamin D
Drug: Vitamin D — Vitamin D administered IV
  Other Names: paricalcitol, doxercalciferol

SUMMARY:
The purpose of this study is to compare the proportion of chronic kidney disease (CKD) subjects on dialysis receiving Sensipar® and low dose vitamin D or escalating doses of vitamin D alone who are able to achieve the National Kidney Foundation-Kidney Disease Outcomes Quality Initiative (NKF-K/DOQI) secondary hyperparathyroidism (HPT) treatment targets for both biointact parathyroid hormone (biPTH) and calcium-phosphorus (Ca x P) product.

ELIGIBILITY:
Inclusion Criteria: - On hemodialysis for at least 3 months and have received intravenous vitamin D therapy (paricalcitol or doxercalciferol) for at least 3 months prior to entering screening - Historical iPTH 150-800 pg/ml (or biPTH 80-430 pg/ml) within 6 months and corrected serum Ca greater than 8.4 mg/dl within 2 months prior to screening period. For subjects with biPTH 80-160 pg/ml (iPTH 150-300 pg/ml), Ca x P must be greater than 55 mg²/dl² within 2 months prior to the screening period - Screening (pre-washout) biPTH 80-430 pg/ml and a corrected serum Ca level greater than 8.4 mg/dl. For subjects with biPTH 80-160 pg/ml Ca x P must be also greater than 55 mg²/dl² - Baseline mean biPTH (post-washout) greater than 160 pg/ml and mean corrected Ca greater than 8.4 mg/dl Exclusion Criteria: - Parathyroidectomy in the 3 month period prior to screening - Current gastrointestinal disorder that may be associated with impaired absorption of orally administered medications or an inability to swallow tablets - Use of investigational drug or device or participation in a trial of investigational drug or device within 30 days of screening - Females of child bearing potential who are pregnant (e.g., positive pregnancy test) or are breast feeding or who refuse to use highly effective contraceptive measures (as determined by the investigator) throughout the study - Previously participated in this or any other Sensipar® study or has received or is receiving Sensipar® as a commercially available product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2005-08; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Achieving the NKF-K/DOQI targets for both biPTH (80-160 pg/mL, equivalent to iPTH 150-300 pg/mL) and Ca x P (less than 55 mg^2/dL^2) during the assessment phase | Weeks 17 - 27
  Proportion of subjects in each treatment group simultaneously achieving the National Kidney Foundation - Kidney Disease Outcome Quality Initiative (NKF-K/DOQI) targets for both biPTH (80-160 pg/mL, equivalent to iPTH 150-300 pg/mL) and Ca x P (< 55 mg^2/dL^2) during the assessment phase (last 11 weeks of study following a 16-week titration phase)

SECONDARY OUTCOMES:
Absolute Change from Baseline for P During the Assessment Phase | Baseline to weeks 17-27
  Absolute change from baseline for serum phosphorus (P) during the assessment phase
Proportion of Participants with ≥ 30% Reduction from Baseline in Mean iPTH During the Assessment Phase | Baseline and Weeks 17-27
  Proportion of participants with ≥ 30% reduction from baseline in mean intact parathyroid hormone (iPTH) during the assessment phase.
Percent Change from Baseline for Calcium During the Assessment Phase | Baseline to weeks 17-27
  Percent Change from Baseline for Calcium (Ca) During the Assessment Phase
Percent Change from Baseline for Phosphorus During the Assessment Phase | Baseline to weeks 17-27
  Percent change from baseline for Phosphorus (P) during the assessment phase
Percent Change from Baseline for Ca x P During the Assessment Phase | Baseline to weeks 17-27
  Percent change from baseline for calcium x phosphorus (Ca x P) during the assessment phase
Percent Change from Baseline for iPTH During the Assessment Phase | Baseline to weeks 17-27
  Percent change from baseline for intact parathyroid hormone (iPTH) during the assessment phase
Proportion of Participants who Attained the K/DOQI Target Range for Ca x P During the Assessment Phase. | Weeks 17 - 27
  Proportion of participants who attained the K/DOQI target range for calcium x phosphorus (Ca x P) during the assessment phase.
Proportion of Participants who Attained the K/DOQI Target Range for Ca During the Assessment Phase | Weeks 17-27
  Proportion of participants who attained the K/DOQI target range for calcium (Ca) during the assessment phase.
Proportion of Participants who Attained the K/DOQI Target Range for iPTH During the Assessment Phase | Weeks 17-27
  Proportion of participants who attained the K/DOQI target range for intact parathyroid hormone (iPTH) during the assessment phase.
Proportion of Participants who Attained the K/DOQI Target Range for P During the Assessment Phase. | Weeks 17-27
  Proportion of participants who attained the K/DOQI target range for phosphorus (P) during the assessment phase.
Absolute Change from Baseline for iPTH During the Assessment Phase | Baseline to weeks 17-27
  Absolute change from baseline for intact parathyroid hormone (iPTH) during the assessment phase.
Absolute Change from Baseline for Ca During the Assessment Phase | Baseline to weeks 17-27
  Absolute change from baseline for calcium (Ca) during the assessment phase
Absolute Change from Baseline for Ca x P During the Assessment Phase | Baseline to weeks 17-27
  Absolute change from baseline for calcium x phosphorus (Ca x P) during the assessment phase.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Fishbane S, Shapiro WB, Corry DB, Vicks SL, Roppolo M, Rappaport K, Ling X, Goodman WG, Turner S, Charytan C. Cinacalcet HCl and concurrent low-dose vitamin D improves treatment of secondary hyperparathyroidism in dialysis patients compared with vitamin D alone: the ACHIEVE study results. Clin J Am Soc Nephrol. 2008 Nov;3(6):1718-25. doi: 10.2215/CJN.01040308. PMID 18945995
- [Background] Shireman TI, Almehmi A, Wetmore JB, Lu J, Pregenzer M, Quarles LD. Economic analysis of cinacalcet in combination with low-dose vitamin D versus flexible-dose vitamin D in treating secondary hyperparathyroidism in hemodialysis patients. Am J Kidney Dis. 2010 Dec;56(6):1108-16. doi: 10.1053/j.ajkd.2010.07.012. Epub 2010 Oct 15. PMID 20951487
- [Background] TBD.Sensipar plus low dose vitamin D (ACHIEVE).Journal-004521;
- [Background] TBD.Time in target.Journal-004521;
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com